CLINICAL TRIAL: NCT07211867
Title: A Digital Intervention to Decrease Self-Stigma Among Pregnant and Postpartum Women With Substance Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202302102; R44DA055161 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-10-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Substance Use Disorder
Keywords: pregnant and postpartum women; self-stigma; digital interventions; substance use disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — elastin microfibril interface located protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhearten with EMI (Experimental): Enhearten is a digital intervention that is designed to foster adherence to medications for addiction treatment (MAT) and treatment retention while considering the unique needs of pregnant and post-partum women, and recently it has been adapted to include features designed to decrease self-stigma among app-users.
  Interventions: Behavioral: Enhearten with EMI
- Waitlist Control Group (Active Comparator): Participants in this arm will have access to the intervention following the trial.
  Interventions: Behavioral: Waitlist Control Group

INTERVENTIONS:
Behavioral: Enhearten with EMI — Enhearten is a digital intervention that is designed to foster adherence to medications for addiction treatment (MAT) and treatment retention while considering the unique needs of pregnant and postpartum women, and recently it has been adapted to include features designed to decrease self-stigma among app-users
  Arms: Enhearten with EMI
Behavioral: Waitlist Control Group — Participants will receive access to Enhearten with EMI following the trial.
  Arms: Waitlist Control Group

SUMMARY:
Digital interventions have the potential to support healthier behaviors among pregnant and postpartum women (PPW) with substance use disorders (SUDs) and may also provide a promising method for reducing their self-stigma. Enhearten is a digital intervention designed to foster adherence to medications for addiction treatment (MAT) while considering the unique needs of PPW, but its effects on self-stigma, treatment retention, and SUD outcomes have not been rigorously tested. The investigators will conduct an individual-level multicenter randomized controlled trial to test the feasibility, acceptability, and efficacy of Enhearten on reducing self-stigma and on improving SUD treatment and recovery outcomes with a stigma-focused ecological momentary intervention (EMI) designed to: 1) screen for feelings of stigma and 2) counteract these vulnerabilities among PPW with SUD via just-in-time interventions.

DETAILED DESCRIPTION:
Pregnant and postpartum women (PPW) with substance use disorders (SUDs) face high levels of self-stigma, the internalization of negative feelings about oneself because of drug misuse. Self-stigma is highly correlated with numerous detrimental consequences including recovery outcomes and reduced engagement with SUD treatment. Furthermore, self-stigma prevents treatment initiation and engagement among PPW with SUDs, leading to additional adverse health outcomes for both mother and baby. Digital interventions have the potential to support healthier behaviors among PPW with SUDs and may also provide a promising method for reducing their self-stigma. Enhearten is a digital intervention that has been enhanced to foster adherence to medications for addiction treatment (MAT) while considering the unique needs of PPW, but its effects on self-stigma, treatment retention, and SUD outcomes have not been rigorously tested. In this study, the investigators will test this augmented version of Enhearten with a stigma-focused ecological momentary intervention (EMI) designed to: 1) screen for feelings of stigma and 2) counteract these vulnerabilities via just-in-time interventions. Specifically, the investigators will conduct an individual-level multi-center randomized control trial (RCT) to test the feasibility, acceptability, and efficacy of Enhearten on reducing self-stigma and on improving SUD treatment and recovery outcomes. Participants will be randomized to one of two groups: Enhearten with EMI or a waitlist control group (i.e., participants will have access to the intervention following the RCT). Recruitment will occur through treatment facilities and recovery homes throughout the United States, referrals from stakeholders including clinicians and peer support specialists, and approved research recruitment registries. This study will determine the efficacy and utility of Enhearten among PPW with SUDs, addressing a promising solution to supplement traditional in-person care, reduce self-stigma, and support continued motivation and adherence to treatment plans along the recovery journey.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and new mothers (up to 12 months postpartum)
* Adult (≥18 years of age)
* Fluent in English
* Currently owns or has ready (daily) access to a smartphone or tablet to use Enhearten.
* Self-reports a history of substance use, excluding alcohol use, nicotine/tobacco use, and drugs taken as prescribed by a physician OR a history of substance use, excluding alcohol use, nicotine/tobacco use, and drugs taken as prescribed by a physician, is identified in chart review as documented by a healthcare provider

Exclusion Criteria:

- Significant cognitive impairment that interferes with their ability to consent and complete study tasks as self-reported or documented in medical charts by a healthcare provider

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Self-stigma about substance use | Baseline through 6-months post-intervention
  Participants in each group will be assessed on levels of perceived self-stigma using the Brief Substance Use Stigma Scale ). The Brief Substance Use Stigma Scale uses a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree". Mean scores will be created with higher scores indicating higher levels of stigma.
Internalized stigma about substance use | Baseline through 6-months post-intervention
  Participants in each group will be assessed on levels of perceived self-stigma using the Internalized Stigma of Substance Abuse Scale (ISSA). The Internalized Stigma of Substance Abuse Scale (ISSA) uses a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". Mean scores will be created with higher scores indicating higher levels of stigma.

SECONDARY OUTCOMES:
Use of Medications for Addiction Treatment (MAT) | Baseline through 6-months post-intervention
  Participants in each group will be assessed on self-reported use of medications for opioid use disorder or other medications for addiction treatment in the past 30 days.
Substance use | Baseline through 6 months post-intervention
  Participants in each group will be assessed on self-reported use of substances for nonmedical purposes (i.e. opioids, methamphetamine, cocaine, MDMAs, etc) in the past 30 days. Substance use and related symptoms will be assessed using modified items from the National Survey on Drug Use and Health (NSDUH).
Substance use cravings | Baseline through 6 months post-intervention
  Participants in each group will be assessed on self-reported cravings to use substances for nonmedical purposes (i.e. opioids, methamphetamine, cocaine, MDMAs, etc). Substance use cravings will be assessed using modified items from the Penn Alcohol Craving Scale (PACS). The scale uses a 0-6 Likert scale for each of its five items, with a total possible score ranging from 0 to 30, where higher total scores reflect more intense or frequent cravings.
Attitudes towards using medication for addiction treatment during pregnancy/postpartum | Baseline through 6 months post-intervention
  Participants in each group will be assessed on an attitudes measure towards use of medications for addiction treatment during the pregnancy/postpartum period, stemming from the Theory of Planned Behavior. This measure uses a 6-point Likert scale ranging from "strongly disagree" to "strongly agree".
Subjective norms towards using medication for addiction treatment | Baseline through 6 months post-intervention
  Participants in each group will be assessed on a subjective norms measure towards use of medications for addiction treatment, stemming from the Theory of Planned Behavior.
Self-efficacy towards using medication for addiction treatment | Baseline through 6 months post-intervention
  Participants in each group will be assessed on a self-efficacy measure towards use of medications for addiction treatment, stemming from the Theory of Planned Behavior.
Mental health symptoms | Baseline through 6 months post-intervention
  Participants in each group will be assessed on symptoms of mental health from the Medical Outcomes Survey, including symptoms related to depression, anxiety, and distress.
Infant feeding intentions | Baseline through 6 months post-intervention
  Participants in each group who are pregnant will be assessed on intent to breastfeed using The Infant Feeding Intentions (IFI) scale. This measure uses a 5-point Likert-type scale ranging from "very much agree" to "very much disagree".
Usability and usefulness of intervention | 1-month post-intervention to 6-months post-intervention
  Participants in the intervention group will be assessed on usability and usefulness of the Enhearten app using a modified version of the Technology Acceptance Model (TAM). The TAM uses a 7-point Likert scale ranging from "totally disagree" to "totally agree" with higher scores indicating higher levels of usability and usefulness.
Acceptability of intervention | 1-month post-intervention to 6-months post-intervention
  Participants in the intervention group will be assessed on acceptability of the Enhearten app using a modified version of the Acceptability of Intervention Measure (AIM) questionnaire. The modified version of the AIM uses a 7-point Likert scale, ranging from "totally disagree" to "totally agree". Mean scores will be created with higher scores indicating higher levels of acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Alex T Ramsey, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The university will share de-identified data from the RCT. Descriptions of study datasets, final codebook and data dictionary, and programming code for data management and analysis will also be made available. Data and documentation will be housed at Washington University but will be made freely available to other investigators who wish to conduct data audits or perform secondary data analyses.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The data will be made available 12 months after trial completion after data cleaning and quality control completion.
Access Criteria: The research team will make datasets available to any individual who makes a direct request to the MPIs and indicates the data will be used for the purposes of research (per CFR Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge"). In sharing participant data, the team will follow Office of Sponsored Projects' data sharing agreements at Washington University in St. Louis.